CLINICAL TRIAL: NCT05831046
Title: Pilot Study for Patient Re-evaluation Software to Improve Emergency Department Waiting Room Congestion
Brief Title: Emergency Department Re-evaluation Software Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00113113
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-01

CONDITIONS: Emergency Department Waiting Room Congestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): Patients who undergo use of the software prior to being re-evaluated by a physician
  Interventions: Other: ED management software
- Healthy Control (No Intervention): Patients undergo care without using the software

INTERVENTIONS:
Other: ED management software — Patients utilize software after being screened, but prior to being re-evaluated by physician
  Arms: Study Arm

SUMMARY:
This is a research study to determine a method in improving emergency department waiting room care by using new software program.

DETAILED DESCRIPTION:
This is a pilot study to determine the effectiveness of an emergency department re-evaluation software, to improve patient flow through an emergency department. The end goal of the study is to provide proof of the efficacy of the software and provide data such that the software can be improved upon. The study will include ED waiting room patients. The study will involve interaction with the software on a tablet for patients and software on a desktop for providers. The providers utilizing the software will not be considered part of the study, but rather focusing on the outcomes of the patients using the software. Patients will be selected by the provider as available for re-evaluation. Each patient will then be randomized into either a control group (software not used) and a "study" group (software used). Data analysis will be performed in conjunction with clinical statisticians at our institution. The risks of this study are primarily derived from patient privacy concerns, which have been addressed in the risk section.

ELIGIBILITY:
Inclusion:

* Individuals that are 18 and older who have been identified with completed lab work.
* Their primary language must be English to follow the instructions of the study.
* Cognitively sound

Exclusion:

* Minors
* Emergency Severity Index (ESI) class 1 patients
* Individual who cannot legally give consent
* Pregnant patients
* Non-english speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Change in LBTC (left before treatment complete) rates | Baseline, up to 1 year
  The primary objective of this study is to determine efficacy of the designed software, which focuses on the identification and disposition of patients who would otherwise become left before treatment complete (LBTC) patients in the ED waiting room.

SECONDARY OUTCOMES:
Change in disposition time | Baseline, up to 1 year
  This study will also track the total time from study intervention to disposition to determine if utilization of the software decreases disposition time.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Siewny, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital Emergency Department, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No